CLINICAL TRIAL: NCT04979494
Title: Association Between Blood Flow of Super Mesenteric Artery (SMA) and Acute Gastrointestinal Injury (AGI) Using Point-of-care Ultrasound in Critical Care Unit
Brief Title: Association Between SMA Flow and AGI in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Xinchen Wang (Other)
Responsible Party: Sponsor-Investigator, Xinchen Wang, Attending Doctor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: PUMCH-JS-2687
Record Dates: First submitted 2021-05-04; First posted 2021-07-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Gastrointestinal Dysfunction; Critical Illness
Keywords: Regional blood flow; Gastrointestinal dysfunction; Critical care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: ultrasound examination — We conduct abdominal ultrasound examinations for each patient.

SUMMARY:
Acute gastrointestinal injury (AGI) is related to poor outcomes of critically ill patients [1] through many underlying mechanisms [2]. It is also a part of the process of multiple organ dysfunction syndrome (MODS). However, the morbidity of acute gastrointestinal dysfunction in critically ill patients is highly underestimated due to the scarcity of accurate measurement and thus the causes are still unclear.

In this study, investigators are going to apply the technique of point-of-care ultrasound (POCUS) evaluation on the bowel diameters, wall thickness and movement combined with intra-abdominal pressure to determine the occurrence of AGI. The superior mesenteric artery (SMA) blood flow is also evaluated by POCUS to find out the association between SMA blood flow and AGI.

DETAILED DESCRIPTION:
1. Patients are recruited within 24 hours of our surgical ICU admission. The patients are mostly admitted for post-surgery monitor in case of complications due to their baseline health conditions. In some cases, patients are admitted from the emergency room because of severe sickness. Those who are with deep sedation and mechanical ventilation during the first ultrasound evaluation are eligible for the study.
2. Written informed consent was obtained from all patients or next of kin before the recruitment.
3. Information will be collected at enrollment, including demographic characteristics, diagnosis, and so on.
4. There will be two phases of ultrasound evaluation. In Phase One, investigators perform ultrasound evaluation within 24 hours after ICU admission to investigate the SMA blood flow in supine position using POCUS. In Phase Two, starting after the enteral feeding has been initiated, usually within 3 days after the enrollment, ultrasound evaluation on GI function will be performed according to gastrointestinal and urinary tract sonography ultrasound (GUTS) protocol using POCUS. GUTS protocol includes the ultrasound measurement for bowel diameter, bowel wall thickness, peristalsis combined with intra-abdominal pressure(IAP) measured through ureteral catheterization. All measurements would be used to calculate GUTS score to grade the AGI [4].

ELIGIBILITY:
Inclusion Criteria:

1. 18 ~ 80 years old;
2. Under deep sedation (RASS score ≤ -3) with mechanical ventilation at the time of enrollment;
3. Acute Physiology and Chronic Health Evaluation II (APACHE-II) score ≥8.

Exclusion Criteria:

1. Pregnancy;
2. Recent gastrointestinal surgery;
3. History of acute or chronic gastrointestinal dysfunction before ICU admission;
4. Primary or secondary vascular malformation of SMA;
5. Any contraindication to the use of ultrasound evaluation (e.g., abdominal incision).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted into the Department of Critical Care Medicine of Peking Union Medical College Hospital, who were eligible of inclusion criteria, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The occurence of acute gastrointestinal injury | Within 24 hours after the initiation of enteral feeding
  Gastrointestinal and urinary tract sonography ultrasound (GUTS) score will be calculate using a combination bowel diameter in centimeters, bowel wall thickness in centimeters, peristalsis (with or without) using ultrasound, and intra-abdominal pressure in millimeters of mercury measured through urethral tubes[3]. GUTS score is ranging from 0 to 4, and a higher GUTS score means worse gastrointestinal function. A GUTS score more than or equal to 2 is considered as acute gastrointestinal injury(AGI)in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Dawei Liu, MSc., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, China

REFERENCES:
- [Background] Reintam Blaser A, Poeze M, Malbrain ML, Bjorck M, Oudemans-van Straaten HM, Starkopf J; Gastro-Intestinal Failure Trial Group. Gastrointestinal symptoms during the first week of intensive care are associated with poor outcome: a prospective multicentre study. Intensive Care Med. 2013 May;39(5):899-909. doi: 10.1007/s00134-013-2831-1. Epub 2013 Jan 31. PMID 23370829
- [Background] Meng M, Klingensmith NJ, Coopersmith CM. New insights into the gut as the driver of critical illness and organ failure. Curr Opin Crit Care. 2017 Apr;23(2):143-148. doi: 10.1097/MCC.0000000000000386. PMID 28092310
- [Background] Perko MJ, Madsen P, Perko G, Schroeder TV, Secher NH. Mesenteric artery response to head-up tilt-induced central hypovolaemia and hypotension. Clin Physiol. 1997 Sep;17(5):487-96. doi: 10.1046/j.1365-2281.1997.05252.x. PMID 9347197
- [Background] Gao T, Cheng MH, Xi FC, Chen Y, Cao C, Su T, Li WQ, Yu WK. Predictive value of transabdominal intestinal sonography in critically ill patients: a prospective observational study. Crit Care. 2019 Nov 27;23(1):378. doi: 10.1186/s13054-019-2645-9. PMID 31775838